CLINICAL TRIAL: NCT00949299
Title: Effects of Buprenorphine on Ulnar Nerve Motor Block
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough could be recruted
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Stv 2/2009
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2011-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: buprenorphine — intradermal injection

SUMMARY:
Recent reports showed that the opioid buprenorphine is a very potent sodium channel blocker. Buprenorphine not only exerts a strong antinociception, but also a long lasting antihyperalgesic effect. This antihyperalgesic effect is not observed for other clinically employed opioids but is common for local anaesthetics.

The principal aim of the study is to compare the speed of onset and the time of recovery of motor blockage achieved by lidocaine and buprenorphine, respectively. The investigators hypothesize that the blocking capacity of buprenorphine is equal to the one of lidocaine.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age: 18 - 65 years
3. Weight: 50-100kg
4. Height: 155-195cm
5. Signed and dated informed consent
6. Sufficient command of German language

Exclusion Criteria:

1. Contraindications to the class of drugs under study
2. Vulnerable subjects (intellectually or mental impaired)
3. Known hypersensitivity to class of drugs or the investigational product
4. Drug abuse
5. Known peripheral neuropathies
6. Diabetes mellitus
7. Chronic alcohol consumption
8. Congestive heart disease
9. Participants of other studies during study period

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The principal aim of the study is to measure the speed of onset and the time of recovery of motor blockage achieved by lidocaine and buprenorphine | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Maurer, MD, Principal Investigator — Oberarzt Institute of Anesthesiology
Locations (1):
- University Hospital Zurich, Institut of Anaesthesiology, Zurich, Canton of Zurich, Switzerland